CLINICAL TRIAL: NCT02817724
Title: Integral Strategy to Supportive Care in Breast Cancer Patients Through Occupational Therapy and a M-health System: a Randomized Controlled Trial.
Brief Title: Integral Strategy to Supportive Care in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Granada (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, Manuel Arroyo Morales, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI14/01627; PI14/01627 (Other Grant/Funding Number: Spanish Ministry of Economy and Competitiveness, Fondo de Investigación Sanitaria del Instituto de Salud Carlos III); FPU14/01069 (Other Grant/Funding Number: Spanish Ministry of Education)
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; survivor; occupational therapy; mobile applications; Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- m-Health group (Active Comparator): BENECA System: The m-health group will use the BENECA app for 8 weeks.
  Interventions: Device: BENECA System
- Integral Group (Experimental): BENECA System and Supervised-occupational therapy program: The integral groups will use the BENECA app and they will receive a face-to-face occupational therapy rehabilitation program for 8 weeks.
  Interventions: Device: BENECA System; Other: Supervised-occupational therapy program

INTERVENTIONS:
Device: BENECA System — BENECA System is a mobile application whit aims to recover a healthy lifestyle in breast cancer survivors (in terms of energy balance: physical activity and dietary).
Other: Supervised-occupational therapy program — It is a comprehensive program that covers most of the physical, cognitive and emotional needs of these patients after oncology treatment from occupational therapy perspective.
  Arms: Integral Group

SUMMARY:
The purpose of this study is to determine if it is better an integral strategy, with a m-health system, when used in addition to a supervised treatment, versus the use of the m-health system alone, to improve the immediate and long-term Quality of Life of breast cancer survivors.

DETAILED DESCRIPTION:
Background: Technological support using e-health mobile applications (m-health) is a promising strategy to improve the adherence to healthy lifestyles in breast cancer survivors (excess in energy intake or low physical activity are determinants of the risk of recurrence, second cancers and cancer mortality). Moreover, cancer rehabilitation programs supervised by health professionals are needed due to the inherent characteristics of these breast cancer patients. Our main objective is to compare the clinical efficacy of a m-health lifestyle intervention system alone versus an integral strategy to improve Quality of Life (QoL) in breast cancer survivors.

Methods: This therapeutic superiority study will use a two-arm, assessor blinded parallel randomized clinical trial (RCT) design. Women will be eligible if: they are diagnosed of stage I, II or III-A breast cancer; are between 25 and 75 years old; have a Body Mass Index > 25kg/m2; they have basic ability to use mobile apps; they had completed adjuvant therapy except for hormone therapy; and they have some functional shoulder limitations. Participants will be randomized to one of the following groups: integral group will use a mobile application (BENECA APP) and will receive a supervised rehabilitation (8-weeks); m-health group will use the BENECA app for 8-weeks. Study endpoints will be assessed after 8 weeks and 24 weeks. The primary outcome will be QoL measured by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core and breast module. The secondary outcomes: body composition; upper-body functionality (handgrip, Disability of the Arm, Shoulder and Hand questionnaire, goniometry); cognitive function (Wechsler Adult Intelligence Scale, Trial Making Test); anxiety and depression (Hospital Anxiety and Depression Scale); and accelerometer.

Discussion: This study has been designed to seek to address the new needs for support and treatment of breast cancer survivors, reflecting the emerging need to merge new low cost treatment options with much-needed involvement of health professionals in this type of patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I, II or IIIA breast cancer.
* Overweight or obese, according to the Spanish Society for the Study of Obesity.
* Basic ability to use mobile apps or living with someone who has this ability.
* Medical clearance of participants.
* Completion of adjuvant therapy except for hormone therapy.
* Some functional or Range of Motion (ROM) limitations measures by goniometry and the DASH Questionnaire.
* Have signed informed consent.

Exclusion Criteria:

* History of cancer recurrence.
* Chronic disease or orthopedic issues that would interfere with the ability to participate in the rehabilitation program.
* Uncontrolled hypertension (diastolic pressure > 95mm Hg).

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QLQ) | Participants will be followed over 8 weeks.
  The primary outcome will be assessed with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORT QLQ-C30) version 3.0., and with the European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality of Life Questionnaire (EORT QLQ-BR23). Both are the most widely used instruments to measure Quality of Life in cancer patients.

SECONDARY OUTCOMES:
Body mass Index | Participants will be followed over 8 weeks.
  Body mass index, in kg/m2, will be assessed by conducting Dual-energy X-ray absorptiometry (DXA, Discovery densitometer from HOLOGIC, QDR 4500W).
Fat mass | Participants will be followed over 8 weeks.
  % Fat mass will also be assessed by conducting Dual-energy X-ray absorptiometry (DXA, Discovery densitometer from HOLOGIC, QDR 4500W).
Abdominal adipose tissue | Participants will be followed over 8 weeks.
  Abdominal adipose tissue will also be assessed by conducting Dual-energy X-ray absorptiometry (DXA, Discovery densitometer from HOLOGIC, QDR 4500W).
Bone mineral density | Participants will be followed over 8 weeks.
  Bone mineral density (Z-score) will also be assessed by conducting Dual-energy X-ray absorptiometry (DXA, Discovery densitometer from HOLOGIC, QDR 4500W).
Shoulder Range of Motion (ROM) | Participants will be followed over 8 weeks.
  - Shoulder ROM measurements will be obtained using a standard, two-armed goniometer which is described as the clinical gold standard.
Upper Body Functionality | Participants will be followed over 8 weeks.
  The disability of the arm, shoulder and hand (DASH) questionnaire will be used to measure the upper extremity functionality. It includes 30-item disability/symptom scale.
Upper body muscular strength | Participants will be followed over 8 weeks.
  Handgrip: Upper body muscular strength will be determined using digital dynamometer (TKK 5101 Grip-D; Tokyo, Japan. The precision will be 0.1 kg.
Cognitive function: attention | Participants will be followed over 8 weeks.
  The trial making test (TMT) will be used to assess speed for attention, sequencing, mental flexibility, visual search and motion function.
Cognitive function: memory and processing speed | Participants will be followed over 8 weeks.
  Wechsler Adult Intelligence Scale (WAIS IV) will be used to assess working memory and processing speed.
Anxiety and depression | Participants will be followed over 8 weeks.
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess levels of anxiety and depression. It contains 14 items (7 items for each scale) with 4-point likert scale.
Physical activity | Participants will be followed over 8 weeks.
  Participants will be asked to wear an try-axial accelerometer (ActiGraph GT3X+, Pensacola, Florida, US) to record physical activity intensity levels and patterns, as well as sleeping habits.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Arroyo-Morales, PhD, Study Director — Deparment of physiotherapy, Faculty of Health Sciences, University of Granada
Locations (1):
- Faculty of Health Sciences. University of Granada, Granada, Spain

REFERENCES:
- [Derived] Lozano-Lozano M, Galiano-Castillo N, Martin-Martin L, Pace-Bedetti N, Fernandez-Lao C, Arroyo-Morales M, Cantarero-Villanueva I. Monitoring Energy Balance in Breast Cancer Survivors Using a Mobile App: Reliability Study. JMIR Mhealth Uhealth. 2018 Mar 27;6(3):e67. doi: 10.2196/mhealth.9669. PMID 29588273
- [Derived] Lozano-Lozano M, Martin-Martin L, Galiano-Castillo N, Alvarez-Salvago F, Cantarero-Villanueva I, Fernandez-Lao C, Sanchez-Salado C, Arroyo-Morales M. Integral strategy to supportive care in breast cancer survivors through occupational therapy and a m-health system: design of a randomized clinical trial. BMC Med Inform Decis Mak. 2016 Nov 25;16(1):150. doi: 10.1186/s12911-016-0394-0. PMID 27887610